CLINICAL TRIAL: NCT01359709
Title: Effects of Contingency Management and Nicotine Replacement Therapy on Youth Smoking
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Philip Morris USA, Inc. (Industry)
Responsible Party: Principal Investigator, Edythe London, Professor of Psychiatry and Biobehavioral Sciences and Molecular and Medical Pharmacology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ASCC-CM-NRT
Record Dates: First submitted 2011-05-19; First posted 2011-05-25 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Cigarette Smoking Behavior
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency Management (Experimental)
  Interventions: Drug: Nicotine polacrilex
- Noncontingent control (Placebo Comparator)
  Interventions: Drug: Nicotine polacrilex

INTERVENTIONS:
Drug: Nicotine polacrilex — Participants will apply Nicoderm (14 mg) patches everyday during this study.
  Other Names: Nicoderm (14 mg)

SUMMARY:
Cigarette smoking is an important public health concern, and it is most often initiated in adolescence. Despite substantial research on smoking cessation in adults, however, relatively little effort has focused on therapeutic approaches to reduce adolescent smoking.

Behavioral interventions, such as contingency management (CM), and pharmacotherapies, such as nicotine replacement therapy (NRT), each have some efficacy in reducing adolescent smoking, and in adults, combination of behavioral and pharmacological approaches is more effective in reducing smoking than either one alone. Little is known about combining these therapeutic approaches in adolescent smokers, and research in this area has been hindered, in part, by the expense and complexity of large-scale clinical trials of the combined treatments and the relative dearth of a cost-effective laboratory procedure. Developing and validating a laboratory model to evaluate the combined effects of CM and pharmacological adjuncts for adolescent smoking is important because such studies can be conducted more rapidly and efficiently, and could provide information on the optimal conditions (e.g., dose) under which pharmacotherapies might augment the positive effects of CM.

The investigators propose to conduct a randomized, placebo-controlled, double-blind, between-groups, 2-week laboratory study. Participants will be randomly assigned to one of the following four groups: CM+nicotine patches, CM+placebo patches, noncontingent control (NC)+nicotine patches and NC+placebo patches. Fifteen participants will be enrolled in each of the four groups, totaling 60 participants. On day 1, participants will arrive to the laboratory for a 1-h session. During this session, breath carbon monoxide (CO) levels, saliva or urinary cotinine levels will be evaluated. Participants will also complete questionnaires on craving, withdrawal and cigarette dependence. Participants will then receive seven patches, to wear for seven days, one patch daily. Five sessions during the days 8 to 12 will serve as CM or noncontingent sessions, and participants will continue wearing patch daily. On these sessions, breath CO levels will be evaluated, and participants will have opportunity to receive payments based on their CO levels, according to the group assignment. If successful, the proposed study will provide a human laboratory model for use in studies of the combined CM and pharmacological approaches for modifying adolescent smoking behavior.

DETAILED DESCRIPTION:
Nicotine dependence typically emerges during adolescence. As almost 90% of adult smokers begin during adolescence (Campaign for Tobacco Free Kids, 2008), it is critical to develop effective treatments for reducing smoking in adolescents. Despite substantial research in adults, relatively little effort has focused on treatments to reduce adolescent smoking.

Current treatment options for adolescent smoking can be broadly categorized into behavioral and pharmacological approaches. Behavioral treatments, such contingency management, reduce adolescent smoking significantly more than control conditions (Grim Shaw and Stanton, 2006; Sussman et al., 2006). Notably, pharmacotherapies, such as nicotine replacement therapy (NRT) are also safe and efficacious in reducing smoking in adolescents (Upadhyaya et al., 2004; Killen et al., 2004; Hurt et al., 2000; Smith et al., 1996). However, there is limited knowledge regarding the combination of behavioral interventions with pharmacotherapies for reducing adolescent smoking (Hanson et al., 2003; Mollohan et al., 2005).

Combinations of behavioral and pharmacological treatments are more efficacious and cost-effective in reducing smoking in adults than either approach alone (Roving et al., 2009; Reus and Smith, 2008; see review in Ingersoll & Cohen's, 2005). For example, combined treatment with nicotine patches and an "Progressive-Reinforcement Reset" contingency management (CM) paradigm (smokers received escalating monetary rewards according to duration of abstinence) increased abstinence from smoking significantly more than nicotine replacement therapy alone in adults (Shoptaw et al., 2002). Such combination therapy could also be more effective in reducing adolescent smoking than individual treatments. Research efforts in this regard have been hindered, in part, by the expense and complexity of outpatient trials and the relative dearth of a less expensive laboratory procedure assessing adolescent smoking.

Developing and validating a laboratory procedure to evaluate the combined effects of CM and pharmacological adjuncts for adolescent smoking is important because human laboratory studies can be conducted more rapidly and efficiently than clinical trials. Randomized, placebo-controlled clinical trials tend to be costly, lengthy and labor-intensive, and should be reserved for only the most promising medications that show at least some level of efficacy in enhancing CM effectiveness in controlled laboratory conditions. Laboratory studies using adolescent smokers might also identify the optimal conditions (e.g., dose, duration of treatment) under which pharmacotherapies might be expected to be synergistic with CM.

This proposal has one specific aim: to evaluate combined effects of CM and NRT treatments for assessing smoking in adolescents. Such a laboratory paradigm could be useful in evaluating potential pharmacotherapies in augmenting the effects of CM in adolescent smokers. We propose to conduct a proof-of-concept study in which 60 adolescent smokers (ages 13-21) will participate in a randomized, placebo-controlled, double-blind, between-groups, 2-week laboratory study. After intake screening, eligible adolescent smokers will be randomly assigned to one of the following four groups: CM+nicotine patches, CM+placebo patches, noncontingent control (NC)+nicotine patches and NC+placebo patches. Fifteen participants will be enrolled in each of the four groups, totaling 60 participants. Participants will be asked to wear one patch daily for the duration of the study. On day 1, participants will arrive to the laboratory for a 1-h session. During this session, breath carbon monoxide (CO) levels, saliva or urinary cotinine levels will be evaluated. Participants will also complete questionnaires on craving, withdrawal and cigarette dependence. Participants will then receive seven patches, to wear for seven days, one patch daily, beginning that day. Everyday between days 8 to 12, participants will arrive to the laboratory for one hour each, and at the end of the session, they will apply a new patch. Five sessions during the days 8 to 12 will serve as CM or noncontingent sessions. On these sessions, breath CO levels, saliva or urinary cotinine levels will be evaluated, and participants will complete questionnaires on craving, withdrawal and cigarette dependence. On these sessions, participants will have opportunity to receive payments based on their CO levels, according to the group assignment. If successful, the proposed study will provide a human laboratory model for use in studies of the combined CM and pharmacological approaches for modifying adolescent smoking behavior.

ELIGIBILITY:
Inclusion Criteria:

* ages 13-21, inclusive
* English-speaking
* Report daily smoking 10 or less cigarettes
* have smoked for at least 6 months
* Expired breath carbon monoxide (CO) levels 6 or more and Urine cotinine levels >100 ng/ml during intake screening
* Sexually active female subjects will be considered eligible for participation only if they are using a double barrier method of birth control (e.g., diaphragm, intrauterine device, or condom along with spermicide) or hormonal contraceptives (such as prescribed "birth control pills", injections, or a prescribed birth control implant). Such birth control methods should have been used for one month before beginning participation in the research study and continue throughout the study.
* Participants' willingness to quit

Exclusion Criteria:

Pregnancy: We will administer a pregnancy test at each study visit. Female participants who are pregnant will not qualify for study and if found pregnant during the study, they will be excluded from further participation.

Medications and Substances:

Evidence (urine analysis) or self-reported current use of psychotropic medications or substances other than:

* Marijuana
* Alcohol
* Nicotine

Language: Lack of fluency in English Note: If a participant is not a fluent English speaker, the language barrier will interfere with performance of psychological tests and completing questionnaires used in the study. The consent form, all questionnaires, and instructions will be given in English.

Psychiatric Disease:

Current or lifetime diagnosis of an Axis I disorder (according to DSM-IV criteria), except for the following:

* Current or lifetime Marijuana Abuse or dependence
* Current or lifetime Nicotine Dependence
* Current or lifetime Alcohol Abuse or dependence
* ADHD or conduct disorders

Neurological:

* Neurological status that is not within normal limits as determined by a physician and as indicated in self-report.
* have serious cardiovascular disease, including uncontrolled hypertension, coronary artery disease, serious cardiac arrhythmias, vasospastic disease, or angina, due to potential cardiovascular effects of nicotine, as determined via the baseline medical history and physical exam
* have a medical condition that could be made worse by treatment with nicotine, including poorly controlled insulin dependent diabetes, uncontrolled hyperthyroidism, pheochromocytoma, severe oropharyngeal, esophageal, or peptic ulcer disease, or severe renal or hepatic impairment as determined via the baseline medical history and physical exam
* have an allergy to adhesive tape or latex or serious dermatologic disease (excluding minor skin conditions such as mild eczema) due to potential for skin allergy to patch
* if a participant's schedule do not permit to complete the 12-day study, and if he/she can not commit to arrive for the scheduled laboratory sessions.
* have a known allergy to nicotine or any component of the nicotine patches
* be receiving treatment with adenosine, bupropion or varenicline due to potential drug-drug interactions

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | All five days (days 8 to 12)
  Percentage of participants continuously abstinent (breath carbon monoxide ≤ 6 ppm) across all five laboratory sessions in the second week (days 8 to 12) in the contingency management + nicotine replacement therapy (CM+NRT) group versus noncontingent control + nicotine replacement therapy (NC+NRT) group.

SECONDARY OUTCOMES:
Smoking craving (Change from baseline on day 12) | Baseline (day 1), day 12
  The measures used will be: Urge to Smoke (UTS)
Smoking withdrawal (Change from baseline on day 12) | Baseline (day 1), day 12
  The measures used will be: Minnesota Withdrawal Scale (MNWS)
Profile of mood states (Change from baseline on day 12) | Baseline (day 1), day 12
  The measures used will be Profile of Mood States (POMS)
Cigarette dependence (Change from baseline on day 12) | Baseline (day 1), day 12
  The measures used will be: Cigarette Dependence Scale (CDS-12)
Breath carbon monoxide (CO) levels (change from baseline on day 12) | Baseline (day 1), day 12

CONTACTS AND LOCATIONS:
Overall Officials: Edythe D London, Ph.D., Principal Investigator — University California, Los Angeles
Locations (1):
- University California, Los Angeles, Los Angeles, California, United States